CLINICAL TRIAL: NCT04022889
Title: A Randomized, Multi-center, Open-label, Controlled, In Vivo Study to Assess the Recovery and Survival of Radiolabeled Autologous INTERCEPT Apheresis Platelet Components Suspended in 100% Plasma Stored for up to 7 Days
Brief Title: In Vivo Study to Assess the Recovery and Survival of Radiolabeled Autologous INTERCEPT Apheresis Platelet Components Suspended in 100% Plasma Stored for up to 7 Days
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLI 00127
Record Dates: First submitted 2019-07-09; First posted 2019-07-17 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: INTERCEPT; Recovery; Survival; 7 days; Radiolabeled; Autologous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stage 1 (Experimental): The study will be performed in two stages. Stage 1 is a randomized, 2-period crossover design. Test platelets stored for 7 days will be radiolabeled based on either the BEST or Variant 1 methods (depending on the period and randomization scheme for the Test platelets) for 12 healthy subjects. The recovery and survival for Test platelets prepared with the BEST and Variant 1 methods will be compared with each other and against the fresh platelet Control. With agreement from the FDA (BQ200481, July 8, 2020), completion of Stage 1 is not required.
  Interventions: Device: INTERCEPT Treated Platelets
- Stage 2 (Experimental): Stage 2 is a single arm design. Test platelets from 24 healthy subjects, stored for 7 days, will be prepared for radiolabeling following the Variant 1 methodology. The recovery and survival for Test platelets will be compared against the fresh platelet Control. Stage 1 subjects with evaluable Variant 1 method data will contribute to the requirement of the 24 subjects for Stage 2.
  Interventions: Device: INTERCEPT Treated Platelets

INTERVENTIONS:
Device: INTERCEPT Treated Platelets — Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets (Test Platelets) and stored for 7days at 20-24°C with continuous agitation. Samples from the Test component will be processed with either the BEST or the Variant 1 procedure prior to radiolabeling. The radiolabeled autologous Test and Control platelets (approximately 10-30 mL) will be simultaneously administered intravenously into the subject.

SUMMARY:
The principle objective of this study is to evaluate the hypothesis that INTERCEPT Platelets in 100% plasma stored for 5 or more days (up to 7 days) after apheresis collection retain sufficient viability for therapeutic transfusion efficacy. The post-infusion recovery and survival of autologous radiolabeled 7 day INTERCEPT platelets (Test) stored in 100% plasma will be measured in comparison to "fresh" autologous radiolabeled platelets (Control) according to FDA guidance for platelet testing (FDA 1999) in Stage 2 of this study protocol.

A secondary objective is to compare the recovery and survival results for Test platelets prepared for radiolabeling using the procedures outlined by the Biomedical Excellence for Safer Transfusion Collaboration (BEST) or a variation of the BEST procedure (referred to as Variant 1) in Stage 1 of this study protocol. Cerus has demonstrated that the Variant 1 method, which does not incorporate an initial soft spin in the presence of ACD A, results in improved in vitro platelet recovery and quality during preparation for radiolabeling compared to the BEST procedure. This comparison will evaluate the hypothesis that preparation methods prior to radiolabeling may influence in vitro quality of the radiolabeled platelets and post-infusion viability outcomes.

DETAILED DESCRIPTION:
The study will be performed in two stages. Stage 1 is a randomized, 2-period crossover design. Test platelets stored for 7 days will be radiolabeled based on either the BEST or Variant 1 methods (depending on the period and randomization scheme for the Test platelets) for 12 healthy subjects. The recovery and survival for Test platelets prepared with the BEST and Variant 1 methods will be compared with each other and against the fresh platelet Control. With agreement from the FDA (BQ200481, July 8, 2020), completion of Stage 1 is not required.

Stage 2 is a single arm design. Test platelets from 24 healthy subjects, stored for 7 days, will be prepared for radiolabeling following the Variant 1 methodology. The recovery and survival for Test platelets will be compared against the fresh platelet Control. Stage 1 subjects with evaluable Variant 1 method data will contribute to the requirement of the 24 subjects for Stage 2.

For both stages, the study population will consist of healthy subjects who meet the FDA, AABB, and site-specific research donor eligibility criteria for apheresis platelet donation. Apheresis platelets will be collected in 100% plasma on the Trima Accel® Automated Blood Collection system.

Each study apheresis collection will be processed using the INTERCEPT Blood System for Platelets. Platelet components containing 3.0 to 7.9 x10^11 platelets in 300 to 420 mL of plasma will be processed using the INTERCEPT Dual Storage (DS) set. The INTERCEPT process will begin on either the day of collection (Day 0) or the day following donation (Day 1); illumination must occur within 24 hours after the end of collection. Test platelets components will be stored for up to 7 days, from day of collection, in 100% plasma.

During each stage samples for in vitro platelet testing will be collected prior to INTERCEPT treatment (Day 0/1), post INTERCEPT treatment and at the end of storage, Day 7 (see In vitro evaluation of platelets below).

At the end of storage, an aliquot of Test platelets will be aseptically removed from each subject's INTERCEPT platelet storage container for preparation of samples for radiolabeling using either the BEST (Stage 1) or Variant 1 (Stages 1 and 2) methodology. The in vitro quality of the Test platelet sample used for radiolabeling will be assessed prior to and following the pre-radiolabeling platelet sample preparations. The indices to be measured in Stage 1 are volume, pH22°C, CD62P, platelet count, red blood cell (RBC) count and white blood cell (WBC) count. Assessments of these indices will enable the determination of platelet processing recovery for each sample preparation method and evaluation of RBC and WBC contamination in samples prior to radiolabeling. In Stage 2 platelet processing recovery during sample preparation will be calculated from volume and platelet count and pH22°C, will be measured in the sample prior to radiolabeling.

On the day corresponding to the end of storage for the Test component, healthy subjects will return to the site, and 43 mL of whole blood (WB) will be drawn into a syringe containing 9 mL of Anticoagulant Citrate Dextrose Solution, Formula A (ACD A). The sample will be used to prepare Control platelets following the BEST methodology. Test and Control platelets will be randomly radiolabeled with either 51Cr (approximately10-30μCi) as sodium radiochromate (Na251CrO4) or 111In (approximately 10-30 μCi) as indium oxine, depending upon the randomization assignment and period as applicable. Subjects will be randomized with equal probability to the radiolabeling sequences (111In/51Cr vs. 51Cr/111In) for Test/Control. The isotope labels will be assigned randomly with equal probability that Control and Test platelets will be labeled with each isotope, and the same randomization assignment of isotope labels will be utilized for both apheresis collections for the same subject in Stage 1. After radiolabeling, the autologous Control and Test platelet samples will be simultaneously infused into the subject (approximately 10 30 mL). A negative pregnancy test for females of childbearing potential is required before infusion.

Blood samples will be drawn immediately before infusion and for radioactivity measurements at 1 hour ± 15 min and 2 hours ± 15 min post-infusion (Day 0), and 6 more samples will be drawn at 1, 2, 3, 4 (or 5 or 6), 7 or 8, and 11±1 days post-infusion (DPI), at approximately the same time of day as the radiolabeled platelet infusion was administered (±4 hours). The exact time of each sample draw will be recorded.

For subjects enrolled in Stage 1, there will be a minimum washout period of four weeks between the two study periods (e.g., four weeks after the last blood sample at 11±1 DPI, in Period 1). Subjects will be monitored for safety (adverse events) from the first apheresis procedure until 24 hours after the last DPI blood sample is drawn.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years, of either gender.
* Normal health status (as determined by the Investigator review of medical history and blood donor physical exam).
* Meet FDA, AABB, and site guidelines for blood donation and apheresis platelet donation. Travel, tattoos/piercings and/or male to male sexual contact deferrals do not apply.
* Complete blood count (CBC) and serum chemistry values within established reference ranges or within guidelines as above.
* Pre-donation platelet count of more than 150×10^9 platelets/ L.
* Negative blood donor screening test panel for HIV, HBV, HCV, HTLV, syphilis, and WNV.
* Subjects of childbearing potential must agree to use a medically acceptable method of contraception throughout the study. A barrier method of contraception must be included, regardless of other methods.
* Signed and dated informed consent form.

Exclusion Criteria:

* For participation in Stage 2, received any previous infusion in this study.
* Clinically significant acute or chronic disease (as determined by the Investigator).
* Pregnant or nursing females.
* Subjects of childbearing potential not using effective contraception.
* Disease states or conditions that preclude apheresis platelet donation per AABB reference standards.
* Treatment with aspirin or aspirin-containing medications within 7 days of apheresis or treatment with non-steroidal anti-inflammatory drugs (NSAID), anti-platelet agents (or other drugs affecting platelet viability within 3 days of apheresis (e.g., ibuprofen or other NSAIDs).
* Subject received platelet inhibitors within 14 days of donation (e.g., clopidogrel, ticlopidine, amphetamines (e.g., Adderall, Dexedrine)).
* Subjects with positive cocaine and/or amphetamine results from urine drug screen.
* Splenectomized subjects.
* History of known hypersensitivity to indium or chromium.
* Has received an investigational drug within the past 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Bloodworks Northwest Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A subject was considered "enrolled" upon signing the informed consent form.
Pre-assignment Details: Subjects who initiated an apheresis collection were included in the Safety Analysis Set. Subjects with paired Test and Control in vivo recovery and survival data were included in the Evaluable Analysis Set. Data from subjects who completed a Variant 1 arm of Stage 1 was included as part of the Stage 2 analysis.
Groups:
- Stage 1- BEST - Variant 1; Stage 1- Variant 1 BEST: Stage 1 is a randomized, 2-period crossover design. Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) stored for 7 days were radiolabeled based on either the BEST or Variant 1 methods (depending on the period and randomization scheme for the Test platelets) for 12 healthy subjects.
  A subject was considered "enrolled" upon signing the informed consent form. The Safety Analysis Set comprised all subjects who initiated an apheresis collection.
- Stage 2-Variant 1: Stage 2 was a single arm design. Test (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) platelets stored for 7 days, were prepared for radiolabeling following the Variant 1 methodology. The recovery and survival for Test platelets was compared against the fresh platelet Control. A subject was considered "enrolled" upon signing the informed consent form. The Safety Analysis Set comprised all subjects who initiated an apheresis collection. Stage 1 subjects with evaluable Variant 1 method data contributed to Stage 2.
Period: Stage 1: Period 1
Arm/Group | Stage 1- BEST - Variant 1 | Stage 1- Variant 1 BEST | Stage 2-Variant 1
Started (Consented Subjects) | 9 | 6 | 0
Met Screening Criteria | 9 | 6 | 0
Successful Apheresis Collection | 8 | 6 | 0
Completed 7-days Storage of Test Platelet Component | 7 | 6 | 0
Completed Post Infusion Sampling | 7 | 6 | 0
Completed | 7 | 6 | 0
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Platelet component did not meet input specifications | 1 | 0 | 0
Period: Stage 1: Period 2
Arm/Group | Stage 1- BEST - Variant 1 | Stage 1- Variant 1 BEST | Stage 2-Variant 1
Started | 7 | 6 | 0
Met Screening Criteria | 7 | 6 | 0
Successful Apheresis Collection | 7 | 6 | 0
Completed 7-days Storage of Test Platelet Component | 7 | 6 | 0
Completed Post Infusion Sampling | 6 | 5 | 0
Completed | 6 | 5 | 0
Not Completed | 1 | 1 | 0
Not completed — Site closure due to COVID-19 pandemic | 1 | 1 | 0
Period: Stage 2
Arm/Group | Stage 1- BEST - Variant 1 | Stage 1- Variant 1 BEST | Stage 2-Variant 1
Started | 7 (Subjects with Stage 1 Variant 1 data that was included in Stage 2 analysis) | 6 (Subjects with Stage 1 Variant 1 data that was included in Stage 2 analysis) | 22 (Includes only subjects enrolled during Stage 2)
Met Screening Criteria | 7 | 6 | 19
Successful Apheresis Collection | 7 | 6 | 15
Completed 7-days Storage of Test Platelet Component | 7 | 6 | 14
Completed Post Infusion Sampling | 6 | 6 | 14
Completed | 6 | 6 | 14 (Data from 3 completed subjects was not evaluable due to a protocol deviation)
Not Completed | 1 | 0 | 8
Not completed — Screen Failure | 0 | 0 | 3
Not completed — Ineligible for apheresis donation | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Site closure due to COVID-19 pandemic | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A subject was considered "enrolled" upon signing the informed consent form. Safety Analysis Set which was comprised all subjects who initiated an apheresis collection. There were 15 subjects in the Safety Analysis set for Stage 1. The Safety Analysis Set for Stage 2 was comprised on 12 Stage 1 subjects with evaluable Variant 1 method data and 17 new Stage 2 subjects. The demographics for Stage 2 are only for the 17 new Stage 2 subjects.
Groups:
- Stage 1: Stage 1 was comprised of a randomized 2-arm, 2-period crossover design (Period 1 and Period 2). Each subject was randomized to Arm 1 or 2 of the study to determine which methodology was used in Period 1 and Period 2 to prepare and radiolabel the Test platelets. In Arm 1, Test platelets were radiolabeled using the Variant 1 method in Period 1 and the BEST method in Period 2. Test platelets in Arm 2 were radiolabeled using the BEST method in Period 1 and the Variant 1 method in Period 2.
  Test platelets were derived from apheresis platelet components in 100% plasma, collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets and stored for 7 days.
  The recovery and survival for Test platelets was compared against the fresh platelet Control.
  A subject was considered "enrolled" upon signing the informed consent form. Demographics are summarized for the Safety Analysis Set which was comprised all subjects who initiated an apheresis collection for Stage 1.
- Stage 2: Stage 2 was comprised of a single period. Test platelets were derived from apheresis platelet components in 100% plasma, collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets and stored for 7 days. On Day 7 Test platelets were prepared for radiolabeling following the Variant 1 methodology. The recovery and survival for Test platelets was compared against the fresh platelet Control. A subject was considered "enrolled" upon signing the informed consent form. Safety Analysis Set which comprised all subjects who initiated an apheresis collection; the Safety Analysis Set for Stage 2 comprised 12 Stage 1 subjects with evaluable Variant 1 method data and 17 new Stage 2 subjects. Demographics are summarized for the 17 new Stage 2 subjects.
- Total: Total of all reporting groups
Arm/Group | Stage 1 | Stage 2 | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (14.2) | 40.9 (16.2) | 38.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 15 | 29
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32
Height [Mean (Standard Deviation); unit: cm] | 180 (8) | 172 (7) | 176 (8)
Weight [Mean (Standard Deviation); unit: kg] | 93 (16) | 85 (16) | 88 (15)
Blood Type [Number; unit: participants]
  A | 7 | 6 | 13
  B | 2 | 0 | 2
  O | 6 | 10 | 16
  AB | 0 | 1 | 1
Rh Factor [Number; unit: participants]
  Negative | 3 | 2 | 5
  Positive | 12 | 15 | 27
BMI [Mean (Full Range); unit: kg/m^2] | 29 [21 to 43] | 29 [20 to 44] | 29 [20 to 44]

OUTCOME MEASURES:

1. Primary Outcome: Post Infusion Recovery of Test Platelets at End of Storage (Day 7)
Description: Recovery of Test platelets stored for 7 Days as compared to fresh controls. In vivo recovery was expressed as proportion of infused in days and was estimated using a multiple-hit model. The FDA acceptance criteria for survival is >66% of control with the lower bound of a two-sided 95% CI for the mean treatment difference (Test-0.66*Control) in survival is greater than or equal to zero.
Time Frame: 11 days (+/- 1 day) post infusion of radiolabeled Test platelets stored for 7 days and fresh Control platelets
Population: The Evaluable Analysis Set (EAS) comprised all infused subjects who had both paired (referred to Test and Control) recovery and paired survival data for the relevant study stage and/or radiolabeling method, and otherwise complied with the protocol without any other major protocol deviation. EAS was the primary analysis population for the efficacy evaluation.
Measure: Mean (Standard Deviation); unit: percentage of infused platelets
Groups:
- Stage 1 - Variant 1 Arm - TEST: Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) stored for 7 days were radiolabeled with Variant 1 method.
- Stage 1 - Variant 1 Arm - CONTROL; Stage 1 - BEST Arm - CONTROL: An aliquot of autologous, freshly prepared platelets derived from a whole blood sample, collected on the day of infusion and radiolabeled based on the BEST method.
- Stage 1 - BEST Arm- TEST: Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) stored for 7 days were radiolabeled based on the BEST method.
- Stage 2 - TEST: Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) stored for 7 days were radiolabeled with Variant 1 method. Twelve Stage 1 subjects with evaluable Variant 1 method data contributed to Stage 2.
- Stage 2 - CONTROL: An aliquot of autologous, freshly prepared platelets derived from a whole blood sample, collected on the day of infusion and radiolabeled based on the BEST method. Twelve Stage 1 subjects with evaluable Variant 1 method data contributed to Stage 2.
Arm/Group | Stage 1 - Variant 1 Arm - TEST | Stage 1 - Variant 1 Arm - CONTROL | Stage 1 - BEST Arm- TEST | Stage 1 - BEST Arm - CONTROL | Stage 2 - TEST | Stage 2 - CONTROL
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 23 | 23
percentage of infused platelets | 39.5 (10.3) | 57.8 (11.6) | 39.1 (10.6) | 60.4 (10.5) | 37.6 (8.4) | 56.8 (9.2)
Statistical Analysis 1: Comparison: Stage 1 - Variant 1 Arm - TEST vs Stage 1 - Variant 1 Arm - CONTROL; Test type: Non-Inferiority — The null hypothesis of inferiority was to be rejected in favor of the alternative hypothesis of non-inferiority at the two-sided 0.05 significance level if the lower bound of a two-sided 95% CI for the mean treatment difference (Test - 0.66 × Control) was greater than or equal to zero; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-3.5 to 6.2], Standard Deviation 7.7 — The mean treatment difference is defined as Test recovery - (0.66 × Control recovery)
Statistical Analysis 2: Comparison: Stage 1 - BEST Arm- TEST vs Stage 1 - BEST Arm - CONTROL; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-6.4 to 4.8], Standard Deviation 8.9 — The mean treatment difference is defined as Test recovery - (0.66 × Control recovery)
Statistical Analysis 3: Comparison: Stage 1 - Variant 1 Arm - TEST vs Stage 1 - BEST Arm- TEST; Test type: Other — Variant 1-BEST = Test Variant 1 Endpoint - Test BEST Endpoint; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-5.0 to 8.7], Standard Deviation 10.2 — The mean treatment difference is defined as Test recovery - (0.66 × Control recovery)
Statistical Analysis 4: Comparison: Stage 2 - TEST vs Stage 2 - CONTROL; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.5 to 2.6], Standard Deviation 5.9 — The mean treatment difference is defined as Test recovery - (0.66 × Control recovery)

2. Primary Outcome: Post Infusion Survival of Test Platelets at End of Storage
Description: Survival of Test platelets stored for 7 Days as compared to fresh controls. In vivo recovery was expressed as proportion of infused in days and was estimated using a multiple-hit model. The FDA acceptance criteria for survival is >58% of control with the lower bound of a two-sided 95% CI for the mean treatment difference (Test - 0.58 * Control) in survival is greater than or equal to zero.
Time Frame: 11 days (+/- 1 day) post infusion of radiolabeled Test platelets stored for 7 days and fresh Control platelets
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Stage 1 - Variant 1 Arm- TEST: Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) stored for 7 days were radiolabeled with Variant 1 method.
Arm/Group | Stage 1 - Variant 1 Arm- TEST | Stage 1 - Variant 1 Arm - CONTROL | Stage 1 - BEST Arm- TEST | Stage 1 - BEST Arm - CONTROL | Stage 2 - TEST | Stage 2 - CONTROL
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 23 | 23
hours | 150.1 (21.6) | 208.9 (15.8) | 143.2 (33.6) | 202.9 (24.4) | 151.4 (20.1) | 209.6 (13.9)
Statistical Analysis 1: Comparison: Stage 1 - Variant 1 Arm- TEST vs Stage 1 - Variant 1 Arm - CONTROL; Test type: Non-Inferiority — The null hypothesis of inferiority was to be rejected in favor of the alternative hypothesis of non-inferiority at the two-sided 0.05 significance level if the lower bound of a two-sided 95% CI for the mean treatment difference (Test - 0.58 × Control) was greater than or equal to zero; Mean Difference (Final Values) = 28.9, 95% CI 2-sided [18.5 to 39.4], Standard Deviation 16.5 — The mean treatment difference is defined as Test survival - (0.58 × Control survival)
Statistical Analysis 2: Comparison: Stage 1 - BEST Arm- TEST vs Stage 1 - BEST Arm - CONTROL; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 25.5, 95% CI 2-sided [9.5 to 41.6], Standard Deviation 25.3 — The mean treatment difference is defined as Test survival - (0.58 × Control survival)
Statistical Analysis 3: Comparison: Stage 1 - Variant 1 Arm- TEST vs Stage 1 - BEST Arm- TEST; Test type: Equivalence — Variant 1-BEST = Test Variant 1 Endpoint - Test BEST Endpoint; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-12.7 to 15.8], Standard Deviation 21.3 — The mean treatment difference is defined as Test survival - (0.58 × Control survival)
Statistical Analysis 4: Comparison: Stage 2 - TEST vs Stage 2 - CONTROL; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 29.8, 95% CI 2-sided [21.8 to 37.8], Standard Deviation 18.5 — The mean treatment difference is defined as Test survival - (0.58 × Control survival)

3. Secondary Outcome: Platelet Dose in Test Component
Description: Percentage of Test components with ≥ 3.0×10^11 platelets
Time Frame: At the end of INTERCEPT treatment on Day 1 or Day 2
Population: Assessed in Test components stored for 7 days for subjects in the Evaluable Analysis Set (comprised all infused subjects who had both paired (referred to Test and Control) recovery and paired survival data for the relevant study stage and/or radiolabeling method, and otherwise complied with the protocol without any other major protocol deviation).
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1 - Variant 1 Arm: Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) stored for 7 days. Samples from this component were radiolabeled with Variant 1 method.
- Stage 1 - BEST Arm: Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) stored for 7 days. Samples from this component were radiolabeled with BEST method.
- Stage 2: Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) stored for 7 days. Samples from this component were radiolabeled with Variant 1 method. Twelve Stage 1 subjects with evaluable Variant 1 method data will contribute to Stage 2.
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
Participants | 12 | 13 | 22

4. Secondary Outcome: Platelet Yield Retention
Description: Percentage of Test components with ≥80% platelet yield retention
Time Frame: At the end of INTERCEPT treatment on Day 1 or Day 2
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
Participants | 12 | 12 | 22

5. Secondary Outcome: pH 22°C
Description: Percentage of Test components with pH 22°C ≥ 6.2
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
Participants | 13 | 13 | 23

6. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Component Volume
Description: Component volume was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
mL | 334 (17) | 338 (12) | 330 (20)

7. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Platelet Count
Description: Platelet count was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ×10^3 platelets/µL
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
×10^3 platelets/µL | 1116 (185) | 1086 (112) | 1133 (176)

8. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Platelet Dose
Description: Platelet dose was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ×10^11 platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
×10^11 platelets | 3.7 (0.7) | 3.7 (0.4) | 3.7 (0.5)

9. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: MPV
Description: MPV was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
fL | 7.3 (0.6) | 7.2 (0.7) | 7.0 (0.7)

10. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: pO2
Description: pO2 was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
mm Hg | 152.2 (7.6) | 147.2 (13.8) | 152.3 (8.3)

11. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Normalized pO2
Description: pO2 normalized for platelet count was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µmol/hrs/10^12 platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
µmol/hrs/10^12 platelets | 43.5 (10.6) | 42.4 (7.3) | 42.5 (8.4)

12. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: pCO2
Description: pCO2 was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
mm Hg | 26.5 (3.1) | 27.4 (2.3) | 26.3 (2.8)

13. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Normalized pCO2
Description: pCO2 was normalized for platelet count and summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µmol/hrs/10^12 platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
µmol/hrs/10^12 platelets | 7.4 (1.0) | 7.8 (0.6) | 7.3 (1.3)

14. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: HCO3
Description: HCO3 was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
mmol/L | 7.4 (2.3) | 7.0 (1.7) | 7.1 (2.1)

15. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Normalized HCO3
Description: HCO3 was normalized for platelet count and was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/10^12 platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
mmol/10^12 platelets | 6.8 (2.7) | 6.5 (1.6) | 6.5 (2.5)

16. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Supernatant Glucose
Description: Supernatant glucose was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
mmol/L | 12.0 (2.4) | 12.0 (2.2) | 12.2 (3.9)

17. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Normalized Supernatant Glucose
Description: Supernatant glucose was normalized for platelet count and summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/10^12 platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
mmol/10^12 platelets | 11.3 (4.2) | 11.1 (2.0) | 11.2 (4.4)

18. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Supernatant Lactate
Description: Supernatant lactate was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 22
mmol/L | 11.6 (3.1) | 11.1 (2.8) | 12.3 (2.8)

19. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Normalized Supernatant Lactate
Description: Supernatant lactate was normalized for platelet count and summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/10^12 platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 22
mmol/10^12 platelets | 10.7 (3.4) | 10.4 (3.1) | 11.1 (2.8)

20. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Total ATP
Description: Total ATP was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µmol/dL
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
µmol/dL | 3.5 (2.1) | 3.0 (1.5) | 4.0 (2.0)

21. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Normalized Total ATP
Description: Total ATP was normalized for platelet count and summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/10^8 platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
nmol/10^8 platelets | 3.2 (2.0) | 2.8 (1.5) | 3.5 (1.7)

22. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Morphology
Description: The morphology score quantifies (via phase-contrast light microscopy) the morphological changes of platelets coincident with the full range of platelet activation profile (Units: Kunicki score; Range is 0 to 400). Higher morphology scores represent healthier platelets. Morphology was summarized descriptively for Stage 1 and Stage 2 Test components.
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
score on a scale | 327 (21) | 326 (31) | 324 (22)

23. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Extent of Shape Change
Description: The Extent of Shape Change is a measurement of agonist-induced, disc-to-sphere shape change of platelets using an aggregometer. It is a quantitative assessment of the proportion of platelets that have discoid morphology in a platelet suspension. Higher values indicate better platelet quality. An aggregometer instrument is to make this measurement. Extent of Shape Change was summarized descriptively for Stage 1 and Stage 2 Test components.
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of extent of shape change
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
percentage of extent of shape change | 18.3 (6.7) | 21.5 (8.2) | 16.8 (5.5)

24. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Hypotonic Shock Response
Description: Hypotonic Shock Response is used as an index of platelet integrity and metabolic homeostasis. An aggregometer instrument was used to measure the ability of platelets to recover their volume after being exposed to a hypotonic environment. Higher values of Hypotonic Shock Response indicate better platelet quality. Hypotonic Shock Response was summarized descriptively for Stage 1 and Stage 2 Test components.
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of hypotonic shock response
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
percentage of hypotonic shock response | 45.8 (14.2) | 53.4 (9.1) | 48.6 (16.9)

25. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Supernatant Lactate Dehydrogenase (LDH) Activity
Description: Supernatant levels of LDH in PCs represent normal plasma LDH plus LDH released by platelets through cell leakage and injury. Supernatant LDH activity was summarized descriptively for Stage 1 and Stage 2 Test components.
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
U/L | 238 (70) | 235 (54) | 238 (86)

26. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Normalized Supernatant LDH
Description: Supernatant LDH activity was normalized for platelet count and was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/10^12 platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
U/10^12 platelets | 222 (87) | 220 (62) | 217 (90)

27. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Total LDH Activity
Description: Total LDH activity was normalized for platelet count and was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
U/L | 2278 (458) | 2294 (537) | 2398 (482)

28. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Supernatant LDH Proportion of Total LDH
Description: Supernatant LDH Proportion of Total LDH, ratio of LDH supernatant to the total LDH, was summarized descriptively for Stage 1 and Stage 2 Test components
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of cell free LDH to total LDH
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
percentage of cell free LDH to total LDH | 10.7 (3.1) | 10.6 (3.3) | 10.1 (3.4)

29. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: Baseline Adjusted Lysis
Description: For calculation of baseline adjusted lysis the baseline/input supernatant LDH is subtract from the Day 7 supernatant LDH; the lysis is calculated from from the Day 7 adjusted supernatant LDH and Day 7 total LDH values. Baseline Adjusted Lysis was summarized descriptively for Stage 1 and Stage 2 Test components.
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: - % of cell free LDH increased from base
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
- % of cell free LDH increased from base | 4.7 (2.7) | 4.6 (2.9) | 4.4 (2.9)

30. Other Pre Specified Outcome: Assessment of the Stored Test (INTERCEPT) Platelet Components: P-selectin (CD62P)
Description: Measurement of P-selectin (CD62P) exposure is often used as an index of platelet activation as it is translocated from the alpha granule to the plasma membrane during platelet secretion. This is a sensitive assay to quantify platelet potential for activation. Higher levels of P-selectin indicate more activation. P-selectin was measured by flow cytometry and was summarized descriptively for Stage 1 and Stage 2 Test components.
Time Frame: At the end of storage on Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of CD62P platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
percentage of CD62P platelets | 44.7 (19.4) | 45.3 (18.2) | 52.2 (16.5)

31. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: Sample Volume From Component
Description: Stage 1 and Stage 2 sample volume from platelet component was summarized descriptively for Test samples processed using both the BEST (Stage 1) and Variant 1 (Stage 1 and Stage 2) procedures.
Time Frame: Day 7
Population: Assessed in samples from Test components stored for 7 days for subjects in the Evaluable Analysis Set (comprised all infused subjects who had both paired (referred to Test and Control) recovery and paired survival data for the relevant study stage and/or radiolabeling method, and otherwise complied with the protocol without any other major protocol deviation).
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Stage 1 - Variant 1 Arm: Samples from 7-day old Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) prior to addition of radiolabel following Variant 1 method.
- Stage 1 - BEST Arm: Samples from 7-day old Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) prior to addition of radiolabel following BEST method.
- Stage 2: Samples from 7-day old Test platelets (INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets) prior to addition of radiolabel following Variant 1 method. Twelve Stage 1 subjects with evaluable Variant 1 method data will contribute to Stage 2.
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
mL | 46.8 (13.8) | 45.4 (15.4) | 42.9 (14.9)

32. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: Platelet Count
Description: Stage 1 and Stage 2 platelet count was summarized descriptively for Test samples processed using both the BEST (Stage 1) and Variant 1 (Stage 1 and Stage 2) procedures.
Time Frame: Day 7
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ×10^3 platelets/µL
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
×10^3 platelets/µL | 5368 (868) | 3938 (856) | 5265 (1128)

33. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: Platelet Yield (Physical Recovery)
Description: In vitro physical platelet recovery is expressed as the percentage of platelets that are remaining after preparation of the Test sample for radiolabeling, prior to addition of the radiolabel, compared to the number of platelets that were present prior to sample preparation. This measurement shows the loss of platelets during the sample preparations and also provides a process control parameter to ensure that the platelet sample used for radiolabeling is representative of the platelet population in the entire platelet component. Stage 1 and Stage 2 Platelet Yield (Physical Recovery) was summarized descriptively for Test samples processed using both the BEST (Stage 1) and Variant 1 (Stage 1 and Stage 2) procedures.
Time Frame: Day 7
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: percentage of physical recovery
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
percentage of physical recovery | 85.2 (6.8) | 67.7 (12.2) | 84.4 (6.8)

34. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: Percentage of Samples With Physical Recovery ≥ 80%
Description: The percentage of Stage 1 and Stage 2 samples with physical recovery ≥ 80% was summarized for Test samples processed using both the BEST (Stage 1) and Variant 1 (Stage 1 and Stage 2) procedures.
Time Frame: Day 7
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 12 | 23
Participants | 11 | 1 | 16

35. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: pH 22°C
Description: Stage 1 and Stage 2 pH 22°C was summarized descriptively for Test samples processed using both the BEST (Stage 1) and Variant 1 (Stage 1 and Stage 2) procedures.
Time Frame: Day 7
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: pH unit
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
pH unit | 6.3 (0.3) | 6.1 (0.4) | 6.3 (0.2)

36. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: Percentage of Samples With pH 22°C ≥ 6.2
Description: The percentage of Stage 1 and Stage 2 samples with pH 22°C ≥ 6.2 was summarized for Test samples processed using both the BEST (Stage 1) and Variant 1 (Stage 1 and Stage 2) procedures.
Time Frame: Day 7
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm | Stage 2
Number analyzed (Participants) | 13 | 13 | 23
Participants | 8 | 8 | 18

37. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: Red Blood Cell Total Count
Description: The Red Blood Cell Total Count was summarized descriptively for Test samples processed using both the BEST and Variant 1 procedures in Stage 1.
Time Frame: Day 7
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm
Number analyzed (Participants) | 13 | 12
cells | 212 (456) | 176 (324)

38. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: White Blood Cell Total Count
Description: The White Blood Cell Total Count was summarized descriptively for Test samples processed using both the BEST and Variant 1 procedures in Stage 1.
Time Frame: Day 7
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm
Number analyzed (Participants) | 13 | 12
cells | 2666 (3104) | 722 (629)

39. Other Pre Specified Outcome: In Vitro Evaluation of Processed Platelet Samples Prior to Radiolabeling: P-selectin Expression (CD62P)
Description: Measurement of P-selectin (CD62P) exposure is often used as an index of platelet activation as it is translocated from the alpha granule to the plasma membrane during platelet secretion. This is a sensitive assay to quantify platelet potential for activation. Higher levels of P-selectin indicate more activation. Measurement of P-selectin prior to radiolabeling allows assessment of the amount of platelet activation induced by the sample preparation process when compared to the Day 7 P-selectin levels in the platelet component. The P-selectin expression (CD62P) was summarized descriptively for Test samples processed using both the BEST and Variant 1 procedures in Stage 1.
Time Frame: Day 7
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: percentage of CD62P platelets
Arm/Group | Stage 1 - Variant 1 Arm | Stage 1 - BEST Arm
Number analyzed (Participants) | 13 | 13
percentage of CD62P platelets | 54.2 (21.5) | 67.2 (17.7)

ADVERSE EVENTS:
Time Frame: All AE/SAEs that occur following the start of the apheresis collection through 24 hours and from Day 1 to Day 11 ±1post infusion blood sample (1-3 weeks post collection), in both arms of Stage 1 (Variant 1 or BEST) and/or Stage 2. AEs were collected for the Safety Analysis Set, comprised of all subjects who initiated an apheresis collection.
Description: An AE is any untoward medical occurrence in a subject or clinical investigation subject administered an investigational product and which does not necessarily have a causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product whether or not related to the investigational product.
Groups:
- Stage 1-Variant 1; Stage 1-BEST: The study was performed in two stages. Stage 1 was a randomized, 2-period crossover design. Test platelets stored for 7 days were radiolabeled based on either the BEST or Variant 1 methods (depending on the period and randomization scheme for the Test platelets) for 12 healthy subjects. The recovery and survival for Test platelets prepared with the BEST and Variant 1 methods was compared with each other and against the fresh platelet Control. With agreement from the FDA (BQ200481, July 8, 2020), completion of Stage 1 was not required.
  INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets (Test Platelets) and stored for 7days at 20-24°C with continuous agitation. Samples from the Test component were processed with either the BEST or the Variant 1 procedure prior to radiolabeling. The radiolabeled autologous Test and Control platelets (approximately 10-30 mL) was simultaneously administered intravenously into the subject.
- Stage 2-Variant 1: Stage 2 is a single arm design. Test platelets from 23 healthy subjects, stored for 7 days, were prepared for radiolabeling following the Variant 1 methodology. The recovery and survival for Test platelets were compared against the fresh platelet Control. Twelve Stage 1 subjects with evaluable Variant 1 method data contributed to the requirement of the 23 subjects for Stage 2. Stage 2 AEs did not include the Variant 1 subjects from Stage 1.
  INTERCEPT Treated Platelets: Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets (Test Platelets) and stored for 7 days at 20-24°C with continuous agitation. Samples from the Test component were processed with either the BEST or the Variant 1 procedure prior to radiolabeling. The radiolabeled autologous Test and Control platelets (approximately 10-30 mL) were simultaneously administered intravenously into the subject.
Arm/Group | Stage 1-Variant 1 | Stage 1-BEST | Stage 2-Variant 1
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 8/13 | 11/15 | 10/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1-Variant 1 (N=13) | Stage 1-BEST (N=15) | Stage 2-Variant 1 (N=17)
Abdominal distention (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 2 | 1 | 8
Fatigue (General disorders) | 0 | 1 | 0
Injection site extravasation (General disorders) | 1 | 3 | 2
Injection site haematoma (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Vessel puncture site bruise (General disorders) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthraigia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 3 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sites cannot independently publish data from their site until the combined data from all sites has been published. Cerus must review the proposed publication prior to submission to determine if it contains confidential information.

DOCUMENTS (2):
  • Study Protocol (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04022889/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT04022889/SAP_001.pdf